CLINICAL TRIAL: NCT00908778
Title: A Phase 3 Safety and Efficacy Study of Vitreosolve® for Four Ophthalmic Intravitreal Injections For Inducing Posterior Vitreous Detachment in Retinopathy Patients.
Brief Title: A Safety and Efficacy Study of Vitreosolve® for Non-Proliferative Diabetic Retinopathy Subjects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitreoretinal Technologies, Inc. (Industry)
Responsible Party: Hampar Karageozian, CEO
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: PVD- 302
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitreosolve I (Experimental): Intravitreal injection
  Interventions: Drug: Vitreosolve
- Vitreosolve (Experimental): Intravitreal injection
  Interventions: Drug: Vitreosolve

INTERVENTIONS:
Drug: Vitreosolve — intravitreal injection
  Arms: Vitreosolve I
Drug: Vitreosolve — intravitreal injection
  Arms: Vitreosolve

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Vitreosolve® in diabetic retinopathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of systemic diabetes(type I,or II)
* Subject with a documented history of Non- proliferative Diabetic Retinopathy(NPDR)
* Subjects with no or partial PVD at baseline exam in study eye.

Exclusion Criteria:

* Subjects with retinal pathology in the study eye other then (NPDR)
* Subjects with high myopia in the study eye
* Subjects who have monocular vision or central lateral vision of 20/200 or worse BCVA in the non-study eye.
* Subjects with an aphakic study eye or if pseudophakic, cataract extraction surgery less then 6 months prior to study enrollment.
* Subjects that have either vitrectomy surgery, intavitreal injections, or laser treatments in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Ultrasound, OCT, and clinical exam | 6 months

SECONDARY OUTCOMES:
Ultrasound ,OCT ,Safety, and Clinical Exam | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Principal Investigator — APEC, Hospital La Ceguera; Naresh Mandova, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- India (2):
  - LVPEI, Vizag, Andhra Pradesh
  - Amrita, Kochi
- Mexico (3):
  - La Ceguera, San Lucas, Coyoacan
  - Conde De Valenciana, Mexico City, Mexico City
  - Hidalgo, Monterrey, Neuvo Leon